CLINICAL TRIAL: NCT02543411
Title: Effect of Intravenous Lidocaine During Endoscopic Submucosal Dissection for Gastric Neoplasm
Brief Title: Use of Lidocaine in Endoscopic Submucosal Dissection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Severance Hospital (Other)
Responsible Party: Principal Investigator, So Yeon Kim, Assistant professor, Severance Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 4-2014-0933
Record Dates: First submitted 2015-09-02; First posted 2015-09-07 (Estimated); Last update posted 2015-12-15 (Estimated); Status verified 2015-12

CONDITIONS: Gastric Neoplasm
MeSH Terms: conditions — Stomach Neoplasms | interventions — Lidocaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lidocaine group (Experimental): Administration of lidocaine 1%
  Interventions: Drug: Lidocaine 1%
- Control group (Placebo Comparator): Administration of normal saline
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Lidocaine 1% — Intravenous administration as bolus of lidocaine 1.5 mg/kg before sedation and infusion of lidocaine 2 mg/kg/hr during sedation.
  Sedation with fentanyl and propofol
  Arms: Lidocaine group
Drug: Normal saline — Intravenous administration as bolus of normal saline 0.15 mL/kg before sedation and infusion of normal saline 0.2 mL/kg/hr during sedation.
  Sedation with fentanyl and propofol
  Arms: Control group

SUMMARY:
The primary purpose of this study is to investigate the effects of lidocaine on the total administered dose of fentanyl during sedation for endoscopic mucosal resection.

The secondary purpose of this study is to investigate the effects of lidocaine on pain score related with endoscopic mucosal resection at time of 30 min, 6 hr, and 24 hr after procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Endoscopic submucosal dissection for the treatments of early gastric neoplasm

Exclusion Criteria:

1. Allergy to lidocaine
2. Chronic pain
3. Chronic abuse of opioid or NSAID
4. Atrioventricular conductance block
5. Liver dysfunction
6. Renal dysfunction

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2015-09; Primary Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Fentanyl consumption during sedation | During sedation, an expected average of 40 minutes

SECONDARY OUTCOMES:
Pain intensity measured by numerical rating scale | 30 min, 6 hr, and 24 hr after procedure
  0 = no pain at all and 10 = worst pain imaginable (11-point numerical rating scale)
Incidence of nausea and vomiting | Up to 24 hours
  Nausea requiring antiemetics and retching and/or vomiting

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine and Anesthesia and Pain Research Institute, Severance Hospital, Yonsei University College of Medicine, Seoul, South Korea